CLINICAL TRIAL: NCT06775600
Title: Harvest of Human Bone Marrow-Derived Progenitor Cells During Total Hip Arthroplasty for Use in Regenerative Medicine Applications for Blood Vessel and Islet Regeneration.
Brief Title: Stem Cell Isolation From Femoral Heads Post Total Hip Arthroplasty
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: David Hess (Other)
Responsible Party: Sponsor-Investigator, David Hess, Dr. David Hess, Western University, Canada
Organization: Western University, Canada (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 125884
Record Dates: First submitted 2025-01-09; First posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Obesity and Type 2 Diabetes
Keywords: Stem Cell; Diabetes; Obesity; Regeneration
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Type-2 Diabetes (Experimental): Cells are harvested from individuals with Type-2 Diabetes
  Interventions: Procedure: Hip Replacement
- Obesity (Experimental): Cells are Harvested from individuals with obesity
  Interventions: Procedure: Hip Replacement
- Non-Type-2 Diabetic and Non-Obese Controls (Experimental): Cells are harvested from individuals with no Type-2 Diabetes and no Obesity
  Interventions: Procedure: Hip Replacement

INTERVENTIONS:
Procedure: Hip Replacement — Total Hip Arthroplasty where the Femoral Head will be used to harvest stem cells post-extrication from the individual.

SUMMARY:
Femoral heads will be collected at University Hospital (London, ON, Canada) from individuals with type-2 diabetes, obesity, and no T2D/no obesity controls. The femoral head will be taken to the Robarts Research Institute (London, ON, Canada) for lineage-restricted progenitor cell expansion and analyses. There the femoral heads will be used to isolate three stem cell types - Multipotent Stromal Cells, Endothelial Colony Forming Cells, and Hematopoietic Progenitor Cells. The yield and cell surface markers expressed on these cells will be measured using flow cytometry. These cell types will then undergo further analyses of the secretome, tubule forming assays, vascular regenerative cell exhaustion assays, and will be transplanted into immune deficient mice with with femoral artery ligation. These experiments are to assess the differences in function and expression of these cell types between individuals with type-2 diabetes and/or obesity and/or healthy controls.

DETAILED DESCRIPTION:
Femoral Heads will be extracted by Dr. Lanting (Department of Surgery - Division of Orthopaedics) at University Hospital, they will then be transferred to Robarts Research Institute where they will undergo cell isolation and analyses. Multipotent Stromal Cells, Endothelial Colony Forming Cells, and Hematopoietic Progenitor Cells will be extracted from the bone marrow of the femoral heads. These cells will be used to characterize the difference in regenerative progenitor cell number and potential dysfunction in individuals with type 2 diabetes and/or obesity compared to controls. Analysis will include growth kinetics, flow cytometry, Bio Luminescent Imaging and Laser Doppler Perfusion Imaging using a FAL mouse model.

ELIGIBILITY:
Inclusion Criteria:

* Must be 18+ years of age

Exclusion Criteria:

* Diagnosis of bone cancers
* Diagnosis of Rheumatoid arthritis
* Diagnosis of hematopoietic conditions
* Diagnosis of avascular necrosis of the hip
* does not fall within BMI requirements for experimental groups
* Cannot read and/or speak in english

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Cell Yield | Within 24 hours of surgery
  Quantification of how many cells are harvested from each femoral head prior to expansion in vitro
Cellular Growth Kinetics | Time of cell harvest to 8 weeks post harvest
  Quantification of the Growth Kinetics of each cell type during in vitro cell culture post cell harvest.
Cellular Phenotype | Time of cell harvest to 8 weeks post harvest
  Analysis via flow cytometry of the phenotype of each cell type and their respective surface markers that are involved in regenerative pathways.

CONTACTS AND LOCATIONS:
Overall Officials: David A Hess, PhD, Principal Investigator — Western University

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared, unless disseminated in study publication. This is to protect the study participants.